CLINICAL TRIAL: NCT06672536
Title: A Multicenter, Dose-escalation and Dose-expansion, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy Characteristics of SCT520FF in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Multicenter, Phase I/II Study to Evaluate the Safety, Tolerability, PK and Efficacy of SCT520FF in Patients With nAMD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Collaborators: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCT520FF-A201
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: nAMD
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCT520FF dose level 1 treatment (Experimental): SCT520FF dose level 1(0.625mg),IVI,injection once every 4 weeks,three times continuously
  Interventions: Drug: SCT520FF
- SCT520FF dose level 2 treatment (Experimental): SCT520FF dose level 2(1.25mg),IVI,injection once every 4 weeks,three times continuously
  Interventions: Drug: SCT520FF
- SCT520FF dose level 3 treatment (Experimental): SCT520FF dose level 3(2.5mg),IVI,injection once every 4 weeks,three times continuously
  Interventions: Drug: SCT520FF
- eylea 2 mg (Active Comparator): eylea 2 mg,IVI,injection once every 4 weeks,during the study period
  Interventions: Drug: EYLEA 2 MG

INTERVENTIONS:
Drug: SCT520FF — SCT520FF dose level 1，IVI
  Arms: SCT520FF dose level 1 treatment
Drug: SCT520FF — SCT520FF dose level 2，IVI
  Arms: SCT520FF dose level 2 treatment
Drug: SCT520FF — SCT520FF dose level 3，IVI
  Arms: SCT520FF dose level 3 treatment
Drug: EYLEA 2 MG — EYLEA 2 MG,IVI,injection once every 4 weeks,during the study period
  Arms: eylea 2 mg

SUMMARY:
Multicenter, open-label, multi-dose study to evaluate the safety and tolerability in patients with nAMD treated with SCT520FF.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Age≥45 years, ≤80 years，male or femal.
3. The study eye must meet the following criteria: Diagnosis of nAMD;Active MNV lesions secondary to nAMD; Total area of all types of lesions ≤12 optic disc areas; BCVA of the study eye 73~19 letters.

Exclusion Criteria:

1. Macular-related retinal pigment epithelial tears in the study eye; scar, fibrosis, atrophy or dense subfoveal exudation involving the fovea in the study eye.
2. Significant APD or opacity of the refractive medium and miosis in the study eye that affect visual acuity or fundus examination.
3. Aphakia (except intraocular lens) or posterior capsular rupture of the lens in the study eye.
4. The study eye has any eye diseases or medical history other than nAMD that may affect central vision and/or macular examine.
5. MNV caused by non-nAMD exists in the study eye .
6. Active inflammation or infection in either eye before randomization.
7. Known allergy to any component of the study intervention or history of allergy to fluorescein or indocyanine green, any anesthetics or antimicrobial agents used during the course of the study.
8. Abnormal liver and kidney function.
9. Poorly-controlled blood pressure before randomization.
10. History of a cardiovascular and cerebrovascular events, including myocardial infarction, unstable angina pectoris, cerebrovascular accidents (including TIA), other thromboembolic diseases (such as thromboembolic angiitis, etc) within 6 months before randomization.
11. Evidence of significant uncontrolled concomitant diseases.
12. Participated in any drug (other than vitamins and minerals) or device clinical trials within 3 months or the duration of 5 half-lives of the study drug (which is longer) before randomization and have used the test drug or received device treatment.
13. Pregnant, lactating women who can not take contraceptive measures during the trial.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events(TEAE) | From Day 0 up to 196days
  Incidence of treatment emergent adverse events
Treatment-related treatment emergent adverse events(TRAE) | From Day 0 up to 196days
  Incidence of treatment-related treatment emergent adverse events
Serious adverse event(SAE) | From Day 0 up to 196days
  Incidence of serious adverse event
Adverse event of special interest(AESI) | From Day 0 up to 196days
  Incidence of adverse event of special interest
Dose limited toxicity(DLT) | From Day 0 up to 196days
  Incidence of dose-limiting toxicities

SECONDARY OUTCOMES:
Best corrected visual acuity(BCVA) | Day 0 up to 196 days
  Mean change from baseline in BCVA
central retina thickness(CRT) | Day 0 up to 196days
  Mean change from baseline in CRT
PK profile | Day 0 up to 196days
  Change of SCT520FF drug concentration in the blood with time
Cmax | Day 0 up to 196days
  The maximum blood concentration after SCT520FF drug enters the bloodstream
Tmax | Day 0 up to 196days
  Time to the Maximum Concentration of SCT520FF
PD profile | Day 0 up to 196 days
  Detection of free VEGF concentration
Immunogenicity | Day 0 up to 196days
  Positive rate of ADA and NAb

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjing, China